CLINICAL TRIAL: NCT07234461
Title: Sexual Well-being of Women Undergoing Mastectomy and Reconstruction: a National Survey.
Brief Title: Sexual Well-being of Women Undergoing Mastectomy and Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UID 4897; L2-367 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Mastectomy and Breast Reconstruction; Sexual Wellness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey (Experimental): At 1-year follow-up, breast cancer patients who underwent mastectomy and reconstruction are asked to complete several questionnaires after the medical consultation collecting sociodemographic information and their sexual well-being.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — Questionnaires collecting sociodemographic information and their sexual well-being.

SUMMARY:
The study plans to collect data from patients on sexual well-being after mastectomy and immediate reconstruction by surveys.

This data can support preoperative patient counselling and the prevention and care of adverse effects of cancer treatments.

Specific subpopulations of mastectomy women showing severe sexual impairment can be outlined; they may benefit from lifestyle changes and intervention strategies (intravaginal use of diazepam, local hyaluronic acid, intravaginal use of spermidine, pelvic floor gymnastic and physiotherapy).

Our goal is to improve quality of life of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mastectomy for primary breast cancer;
* High-risk healthy patients undergoing risk reducing mastectomies;
* Unilateral and/or bilateral mastectomies;
* If unilateral mastectomy, both patients requiring or not contralateral mammaplasty of the healthy breast;
* All reconstructive procedures included (autologous and heterologous reconstructions).

Exclusion Criteria:

* Patients undergoing breast conservation;
* Patients who previously underwent breast cancer treatment, requiring further surgery for local relapse or secondary breast cancers;
* Delayed post-mastectomy reconstructions;
* Patients not available for e-correspondence.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Sexual well-being | Enrollment visit
  Sexual well-being, a multidimensional construct, will be assessed using a combination of validated and non-validated questionnaires. For each outcome score, descriptive statistics will be reported, including mean, standard deviation, median, and interquartile range. Comparisons of mean scores across predefined subgroups-such as type of reconstruction, systemic and local treatments, menopausal status, obesity, and parity-will be conducted using analysis of variance. A p-value < 0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (19):
- Italy (19):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Italy
  - Istituto Tumori Giovanni Paolo II, Bari, Italy
  - Policlinico Sant'Orsola-Malpighi, Bologna, Italy
  - Ospedale Bufalini di Cesena, Cesena, Italy
  - Presidio Ospedaliero GB Morgagni-Pierantoni, Forlì, Italy
  - European Institute of Oncology, Milan, Italy
  - Ospedale Mater Olbia, Olbia, Italy
  - Azienda Ospedale Università di Padova, Padua, Italy
  - Policlinico Paolo Giaccone, Palermo, Italy
  - Policlinico San Matteo, Pavia, Italy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Italy
  - Campus Biomedico, Roma, Italy
  - Istituto Tumori Regina Elena, Roma, Italy
  - Policlinico Gemelli, Roma, Italy
  - A.O.U. Città della salute e della scienza di Torino, Torino, Italy
  - Azienda Ospedaliera di Treviso, Treviso, Italy
  - Ospedale di Cattinara, Trieste, Italy
  - Ospedale Universitario di Udine, Udine, Italy
  - Breast Unit Settelaghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: No